CLINICAL TRIAL: NCT06814951
Title: Acute Effect of the Thoraco-abdominal Rebalance Method on Diaphragmatic Function, Respiratory Discomfort, Pulmonary Complications and Hemodynamic Variables in Postoperative Cardiac Surgery Patients: Randomized Clinical Trial
Brief Title: Acute Effect of the Thoraco-abdominal Rebalance Method on Diaphragmatic Function, Respiratory Discomfort, Pulmonary Complications and Hemodynamic Variables in Postoperative Cardiac Surgery Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 6075/23
Record Dates: First submitted 2025-02-04; First posted 2025-02-07 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Complications; Diaphragmatic Excursion; Pulmonary Spirometry
Keywords: Physiotherapy; Ultrasonography; Cardiology

STUDY DESIGN:
Intervention Model Description: The randomization technique for the proposed interventions will be performed using a computer program (www.random.org) containing the coded distribution. The allocation confidentiality will be guaranteed by a randomization list that will be kept in a remote location, which will prevent the researcher from identifying which intervention will be initiated by each patient. The generation of the sequence of numbers will be performed by a blinded researcher, after selecting the patients according to the inclusion criteria. The sequence of numbers to be used for randomization will be kept confidential until the exact moment of the beginning of the study. The randomization of the subjects in the proposed groups will be done in two blocks, in which the program will randomly distribute each new participant to one of the blocks: conventional physiotherapy group and RTA group.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physiotherapy (Active Comparator): Patients selected for the control group (conventional physiotherapy) will be exposed to respiratory physiotherapy techniques such as vibrocompression, manual passive expiratory therapy, acceleration of expiratory flow, fractional inspiration in times, diaphragmatic breaths and aspiration when necessary.
  Interventions: Procedure: Conventional physiotherapy
- TAR Method (Active Comparator): Patients selected for the intervention group will undergo thoracoabdominal rebalancing treatment, such as abdominal and/or ileocostal space supports, inspiratory assistance, release of the shoulder girdle, thoracic balance, release of the pectoralis major and deltoid muscles, along with aspiration, if necessary.
  Interventions: Procedure: TAR Method

INTERVENTIONS:
Procedure: TAR Method — Patients selected for the intervention group will undergo thoracoabdominal rebalancing management such as abdominal supports and/or in the ileocostal space, inspiratory assistance, release of the shoulder girdle, thoracic balance, release of the pectoralis major and deltoid muscles together with aspiration if necessary.
  Arms: TAR Method
Procedure: Conventional physiotherapy — Patients selected for the control group (conventional physiotherapy) will be exposed to respiratory physiotherapy techniques such as vibrocompression, manual passive expiratory therapy, acceleration of expiratory flow, fractional inspiration in times, diaphragmatic breaths and aspiration when necessary.
  Arms: Conventional physiotherapy

SUMMARY:
Introduction: The thoracoabdominal rebalancing (TAR) method aims to promote diaphragmatic juxtaposition, in addition to seeking to increase respiratory muscle strength and adjust muscle tone. However, scientific publications on this method in heart patients undergoing coronary artery bypass grafting (CABG) are still scarce, justifying the need to carry out this study for information, evaluation, diagnosis and treatment purposes in the health area with an emphasis on cardiology.

Objective: To evaluate whether diaphragmatic ultrasound findings differ between the TAR method and conventional physiotherapy in post-CABG patients.

Methods: This is a randomized, single-blind clinical trial. Adults (>35 years), hemodynamically stable, who underwent CABG (<24 hours) and had a prescription for physiotherapy will be included. Patients will be randomized into two groups: 1) intervention group [IG] - TAR; 2) control group [CG] - standard physiotherapy approach. Interventions will be performed at a single time and the following variables will be collected pre- and post-intervention: heart rate (HR), respiratory rate (RR), peripheral oxygen saturation (SpO2), mean arterial pressure (MAP), diaphragmatic ultrasound (US) to identify possible acute findings in both groups, respiratory distress scale and pulmonary complications scale will be applied at the end of the interventions.

Keywords: Physiotherapy; Cardiology; Ultrasonography

DETAILED DESCRIPTION:
To compare the effect of conventional physiotherapy techniques with the management of thoracoabdominal rebalancing in postoperative patients after myocardial revascularization surgery, carefully evaluating these effects through diaphragm ultrasound and pulmonary spirometry, in addition to variables such as vital signs and respiratory distress scales and pulmonary complications after cardiac surgery. This is a randomized trial in which patients undergoing myocardial revascularization surgery at the Cardiology Institute of Rio Grande do Sul will participate.

Individuals over 35 years of age who underwent myocardial revascularization surgery with prescribed physiotherapy treatment will be included in the study. Patients who were intubated and/or remained on mechanical ventilation for more than twelve hours or who required non-invasive mechanical ventilation before or during the collection period will be excluded.

The study was submitted to the Research Ethics Committee of the Cardiology Institute of Porto Alegre (CEP-ICFUC). All study participants will receive clear explanations about the research, and those who voluntarily agree to participate in the study will sign the informed consent form in two copies, one of which will be made available to the participant and the other to the researchers. Participants will not be paid, nor will they receive any assistance during or after the end of the research (466/12).

The benefits of this research will be in improved conduct that prevents or reduces complications and/or respiratory discomfort, as well as speeding up the patient's recovery, aiming for faster hospital discharge. Patients selected for the control group (conventional physiotherapy) will be exposed to respiratory physiotherapy techniques such as vibrocompression, passive manual expiratory therapy, acceleration of expiratory flow, fractional inspiration in times, diaphragmatic breathing and aspiration when necessary, and patients selected for group intervention will undergo thoracoabdominal rebalancing management such as abdominal supports and/or in the ileocostal space, inspiratory assistance, release of the shoulder girdle, thoracic swing, release of the pectoralis major and deltoid muscles together with aspiration if necessary.

The research presents minimal risks for the participants, which are related to the measurement of hemodynamic variables through the monitor, in addition to the pulmonary spirometry test and diaphragmatic analysis through ultrasound, and/or application of conventional physiotherapy techniques such as vibrocompression, acceleration of expiratory flow, passive manual expiratory therapy that may suggest some discomfort or pain when touching the chest in a sensation of pressure and vibration. Patients undergoing thoracoabdominal rebalancing treatment are expected to have lower scores on the pulmonary complications scale, Downes and Raphaelly respiratory distress scale and, consequently, better diaphragmatic excursion, as well as improvements in other variables.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 35 years of age who undergo coronary artery bypass graft surgery with prescribed physiotherapy treatment will be included in the study.

Exclusion Criteria:

* Patients who are intubated and/or have remained on mechanical ventilation for more than twelve hours, or who require non-invasive mechanical ventilation (NIV) before or during the collection period will be excluded.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic excursion | Immediately before the intervention and within 30 minutes after the intervention
  Increase in measures
Change in the Downes and Raphaelly respiratory distress scale | Immediately before the intervention and within 30 minutes after the intervention
  Points 0-10, where 0 is best and 10 is worst
Pulmonary spirometry | Immediately before the intervention and within 30 minutes after the intervention
  Increase in measurements: CVF (L)
Pulmonary spirometry | Immediately before the intervention and within 30 minutes after the intervention
  Increase in measurements: VEF1 (L)
Pulmonary spirometry | Immediately before the intervention and within 30 minutes after the intervention
  Increase in measurements: PFE (L/s)
Pulmonary spirometry | Immediately before the intervention and within 30 minutes after the intervention
  Increase in measurements: VEF1/CVF (%)

SECONDARY OUTCOMES:
Respiratory rate | Immediately before the intervention and within 30 minutes after the intervention
  Breathing intervals per minute
Peripheral oxygen saturation | Immediately before the intervention and within 30 minutes after the intervention
  SpO2
Mean arterial pressure | Immediately before the intervention and within 30 minutes after the intervention
  mmHg
Lung auscultation assessment | Immediately before the intervention and within 30 minutes after the intervention
  Wheezing, rhonchi or stridor
Heart rate | Immediately before the intervention and within 30 minutes after the intervention
  Beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Instituto de Cardiologia do Rio Grande do Sul, Principal Investigator — Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Brasil
Locations (1):
- Intituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] SANTANA, Pauliane Vieira et al. Ultrassonografia diafragmática: uma revisão de seus aspectos metodológicos e usos clínicos. Jornal Brasileiro de Pneumologia, v. 46, 2020.
- [Background] Hulzebos EH, Van Meeteren NL, De Bie RA, Dagnelie PC, Helders PJ. Prediction of postoperative pulmonary complications on the basis of preoperative risk factors in patients who had undergone coronary artery bypass graft surgery. Phys Ther. 2003 Jan;83(1):8-16. PMID 12495408
- [Background] OLIVEIRA, Miriana Carvalho; SOBRINHO, Cristina Ortiz; ORSINI, Marco. Comparação entre o método Reequilíbrio Toracoabdominal e a fisioterapia respiratória convencional em recém-nascidos com taquipneia transitória: um ensaio clínico randomizado. Fisioterapia Brasil, v. 18, n. 5, p. 598-607, 2018
- [Background] SOARES, Jainy Lima; DE SOUSA, Anderson Moura Bonfim; DA SILVA MEDEIROS, Joelson. Physiotherapy treatment in the pre and postoperative period of cardiac surgery: an integrative review. Revista Ciência & Saberes-Facema, v. 3, n. 3, p. 624-629, 2017.
- [Background] SANTANA, Vilma Maria et al. Health Education for Patients in the Perioperative Period of Cardiovascular Surgery: Experience Report. Brazilian Journal of Health Review, v. 4, n. 2, p. 5559-5571, 2021.
- [Background] 1. BECCARIA, Lucia Marinilza et al. Postoperative complications in patients undergoing cardiac surgery in a teaching hospital. Archives of Health Sciences, v. 22, n. 3, p. 37-41, 2015.